CLINICAL TRIAL: NCT05683522
Title: Comparison of Postoperative Analgesic Efficacy of Combination of Costaclavicular With Superficial Cervical Plexus Block Versus Subomohyoid Plane Block in Patients Undergoing Arthroscopic Shoulder Surgery
Brief Title: Subomohyoid vs Costoclavicular Block in Shoulder Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samsun University (Other)
Responsible Party: Principal Investigator, Serkan Tulgar, Principal Investigator, Samsun University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SamsunO
Record Dates: First submitted 2023-01-04; First posted 2023-01-13 (Actual); Last update posted 2024-05-28 (Actual); Status verified 2024-05

CONDITIONS: Shoulder Pain
Keywords: Arthroscopic shoulder surgery; Postoperative pain management; Subomohyoid Plane Block; Superficial Cervical Plexus Block; Costaclavicular Block
MeSH Terms: conditions — Shoulder Pain | interventions — Cervical Plexus Block

STUDY DESIGN:
Intervention Model Description: There are two models for this study. The first group is subomohyoid plane block group. The second one is combination of costaclavicular with superficial cervical plexus block.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: The patient and the anesthesiologist who performs postoperative pain evaluation will not know the group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sub-omohyoidal Plane Block (Experimental): Patients randomized to receive sub-omohyoid plane block.
  Interventions: Other: Sub-omohyoidal Plane Block
- Costoclavicular Block plus Cervical Plexus Block (Experimental): Patients randomized to receive costoclavicular brachial and cervical plexus block.
  Interventions: Other: Cervical Plexus Block; Other: Costoclavicular Block

INTERVENTIONS:
Other: Sub-omohyoidal Plane Block — The ultrasound guided sub-omohyoidal plane block will be performed. Patients in this group will be given 15 mL of local anesthetic into the interfascial plane under the omohyoid muscle. This block will be performed preoperatively.
  Arms: Sub-omohyoidal Plane Block
Other: Cervical Plexus Block — A cervical plexus block will be applied by applying 10 mL of local anesthetic under ultrasound guidance. This block will be done before the surgery.
  Arms: Costoclavicular Block plus Cervical Plexus Block
Other: Costoclavicular Block — Costoclavicular brachial plexus block will be applied by administering 20 mL of local anesthetic under ultrasound guidance. This block will be performed preoperatively.
  Arms: Costoclavicular Block plus Cervical Plexus Block

SUMMARY:
Postoperative pain is important following arthroscopic shoulder surgery. Postoperative effective pain treatment provides early mobilization and shorter hospital stay.Ultrasound (US)-guided brachial plexus blocks such as interscalen and supraclavicular block are usually performed. Interscalen brachial plexus block is one of the most preferred techniques among these.

Anterior suprascapular nerve block (subomohyoid plane block), which provides superior trunk block, as described by Siegenthaler et al., has been used for analgesia in shoulder arthroscopies because it is far from the neck and phrenic nerve.

Karmakar et al. described the costoclavicular nerve block, which provides blocking of the posterior, medial and lateral cords of the brachial plexus. It has been suggested as an alternative to postoperative analgesia in shoulder arthroscopies and compared with interscalene brachial plexus block.

The aim of this study is to compare the post op analgesic efficacy of both nerve blocks in shoulder arthroscopic surgeries.

DETAILED DESCRIPTION:
Postoperative pain is an important issue in patients underwent arthroscopic shoulder surgery. Pain causes a few problems; discomfortable patients, negative outcomes and longer rehabilitation. Postoperative effective pain treatment provides early mobilization and shorter hospital stay, thus complications due to hospitalization such as infection and thromboembolism may be reduced. Various techniques may be used for postoperative pain treatment. Opioids are one of the most preferred drugs among the analgesic agents. Parenteral opioids are generally performed for patients after surgery. However opioids have undesirable adverse events such as nausea, vomiting, itching, sedation and respiratory depression (opioid-related adverse events).

Various methods may be performed to reduce the use of systemic opioids and for effective pain treatment following arthroscopic shoulder surgery. Ultrasound (US)-guided brachial plexus blocks such as interscalen and supraclavicular block are commonly used. Interscalen brachial plexus block is one of the most preferred techniques among these.

Ultrasound-guided nerve blocks have been used increasingly due to the advantages of ultrasound in anesthesia practice. US-guided subomohyoid and costoclavicular block are techniques that target the brachial plexus, and their use has increased in recent years. Patients will undergo preoperative subomohyoid block as described by Siegenthaler et al. In the other patient group, costoclavicular block will be applied as described by Karmakar et al. Superficial cervical brachial plexus block will also be applied to this group.

There is no study in the literature about the effectiveness of these techniques against each other. The aim of this study was to evaluate the postoperative analgesic efficacy of the subomohyoid plane block and combination of costoclavicular and superficial cervical plexus block after arthroscopic shoulder surgery.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) classification I-II-III
* Scheduled for arthroscopic shoulder surgery under general anesthesia

Exclusion Criteria:

* history of bleeding diathesis,
* receiving anticoagulant treatment,
* known local anesthetics and opioid allergy,
* infection of the skin at the site of the needle puncture,
* pregnancy or lactation,
* patients who do not accept the procedure

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2023-01-13 (Actual); Primary Completion 2024-05-24 (Actual); Study Completion 2024-05-24 (Actual)

PRIMARY OUTCOMES:
24 hours opioid consumption | up to 24 hours
  morphine consumptions for both group will be recorded

SECONDARY OUTCOMES:
Numeric rating scale for postoperative pain intensity | up to 24 hours
  Changes in Numeric Rating Scale (NRS) at rest and on movement will be recorded at intervals. NRS is a unidimensional measure of pain intensity in adults. The NRS is a segmented numeric version of the visual analog scale (VAS) in which a respondent selects
Quality of Recovery (QoR) | Postoperative 24th hour
  The impact of surgical and anesthetic interventions on perioperative quality of life and ability to resume routine life activities will be assessed using the Quality of Recovery (QoR) tool. The QoR-15 scale is a patient-based outcome measure in the form of a 15-item validated questionnaire.
Incidence of hemidiaphragm paralysis at 30 minutes after sub-omohyoid plan or costoclavicular plus cervical plexus block | 30 minutes post injection
  Ultrasound diagnosed hemidiaphragm paralysis

CONTACTS AND LOCATIONS:
Overall Officials: Serkan Tulgar, Principal Investigator — Samsun University Faculty of Medicine, Samsun Training and Research Hospital
Locations (1):
- Samsun University, Samsun, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Price D. Novel ultrasound-guided suprascapular nerve block. Reg Anesth Pain Med. 2012 Nov-Dec;37(6):676-7; author reply 677. doi: 10.1097/AAP.0b013e3182680bfe. No abstract available. PMID 23086351
- [Background] Sondekoppam RV, Lopera-Velasquez LM, Naik L, Ganapathy S. Subscapularis and sub-omohyoid plane blocks: an alternative to peripheral nerve blocks for shoulder analgesia. Br J Anaesth. 2016 Dec;117(6):831-832. doi: 10.1093/bja/aew370. No abstract available. PMID 27956687
- [Background] Aliste J, Bravo D, Layera S, Fernandez D, Jara A, Maccioni C, Infante C, Finlayson RJ, Tran DQ. Randomized comparison between interscalene and costoclavicular blocks for arthroscopic shoulder surgery. Reg Anesth Pain Med. 2019 Jan 11:rapm-2018-100055. doi: 10.1136/rapm-2018-100055. Online ahead of print. PMID 30635497
- [Background] Abdallah FW, Wijeysundera DN, Laupacis A, Brull R, Mocon A, Hussain N, Thorpe KE, Chan VWS. Subomohyoid Anterior Suprascapular Block versus Interscalene Block for Arthroscopic Shoulder Surgery: A Multicenter Randomized Trial. Anesthesiology. 2020 Apr;132(4):839-853. doi: 10.1097/ALN.0000000000003132. PMID 32044802
- [Background] Karmakar MK, Sala-Blanch X, Songthamwat B, Tsui BC. Benefits of the costoclavicular space for ultrasound-guided infraclavicular brachial plexus block: description of a costoclavicular approach. Reg Anesth Pain Med. 2015 May-Jun;40(3):287-8. doi: 10.1097/AAP.0000000000000232. No abstract available. PMID 25899958